CLINICAL TRIAL: NCT07214792
Title: Understanding Perceptions of and Reactions to Different Food Label Designs
Brief Title: Perceptions of and Reactions to Sustainability Menu Label Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00034378; 5R01DK139327-02 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Food Choices
Keywords: Food labeling; Sustainability; Fast Food
MeSH Terms: interventions — Product Labeling

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view a fast-food online ordering menu with one of seven labeling schemes applied: (1) a QR code on all items (control); (2) Low Sustainability labels; (3) Unsustainable labels; (4) Environmental Harm labels; (5) High Environmental Harm labels; (6) High Environmental Cost labels; and (7) numeric environmental cost labels on all items. All fast-food menus will include a selection of main entrée items. The control QR code and numeric environmental cost labels will display labels on all menu items. All other label conditions will apply labels only to items with higher environmental impact as defined by ingredient-level environmental impact estimates based on the Cool Food Pledge Calculator.
  Participants will be asked about a hypothetical intention to purchase an unspecified menu item with the label to which the participant was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (QR) labels (Placebo Comparator): A black label featuring a QR code and white text that reads "SCAN HERE" will be placed beneath all main menu items.
  Interventions: Behavioral: Control (QR) Labels
- Low Sustainability Labels (Experimental): A red icon-plus-text label that reads "LOW SUSTAINABILITY" in white text will be placed beneath menu items with a high environmental impact, defined by ingredient-level environmental impact estimates from the Cool Food Pledge Calculator.
  Labels will include a white globe icon directly preceding the label text.
  Interventions: Behavioral: Low Sustainability Labels
- Unsustainable Labels (Experimental): A red icon-plus-text label that reads "UNSUSTAINABLE" in white text will be placed beneath menu items with a high environmental impact, defined by ingredient-level environmental impact estimates from the Cool Food Pledge Calculator. Labels will include a white globe icon directly preceding the label text.
  Interventions: Behavioral: Unsustainable Labels
- Environmental Harm Labels (Experimental): A red icon-plus-text label that reads "ENVIRONMENTAL HARM" in white text will be placed beneath menu items with a high environmental impact, defined by ingredient-level environmental impact estimates from the Cool Food Pledge Calculator. Labels will include a white globe icon directly preceding the label text.
  Interventions: Behavioral: Environmental Harm Labels
- High Environmental Harm Labels (Experimental): A red icon-plus-text label that reads "HIGH ENVIRONMENTAL HARM" in white text will be placed beneath menu items with a high environmental impact, defined by ingredient-level environmental impact estimates from the Cool Food Pledge Calculator. Labels will include a white globe icon directly preceding the label text.
  Interventions: Behavioral: High Environmental Harm Labels
- High Environmental Cost Labels (Experimental): A red icon-plus-text label that reads "HIGH ENVIRONMENTAL COST" in white text will be placed beneath menu items with a high environmental impact, defined by ingredient-level environmental impact estimates from the Cool Food Pledge Calculator. Labels will include a white triangle icon with a dollar sign directly preceding the label text.
  Interventions: Behavioral: High Environmental Cost Labels
- Numeric Environmental Cost Labels (Experimental): Numeric Environmental Cost labels will be placed beneath all menu items and display the estimated dollar value associated with the item's True Cost Accounting which calculates the additional cost of a commodity by accounting for environmental and social costs. The label will read "ENVIRONMENTAL COST" in white text followed by a dollar value (i.e., +$6.01). All labels have a solid red background and an icon-plus-text design. A white globe icon will precede the text.
  Interventions: Behavioral: Numeric Environmental Cost Labels

INTERVENTIONS:
Behavioral: Control (QR) Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. Control (QR) labels will be displayed beneath each item. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Control (QR) labels
Behavioral: Low Sustainability Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. Low Sustainability labels will be displayed beneath select items. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Low Sustainability Labels
Behavioral: Unsustainable Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. Unsustainable labels will be displayed beneath select items. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Unsustainable Labels
Behavioral: Environmental Harm Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. Environmental Harm labels will be displayed beneath select items. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Environmental Harm Labels
Behavioral: High Environmental Harm Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. High Environmental Harm labels will be displayed beneath select items. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: High Environmental Harm Labels
Behavioral: High Environmental Cost Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. High Environmental Cost labels will be displayed beneath select items. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: High Environmental Cost Labels
Behavioral: Numeric Environmental Cost Labels — Participants will view a fast-food restaurant menu with main entrée items. Each menu item will be displayed with an image of the item, name, price, and total calories. Numeric environmental cost labels will be displayed beneath each item. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Numeric Environmental Cost Labels

SUMMARY:
The primary objective of this study is to explore perceptions and understanding of different menu label designs related to sustainability and environmental harm. Participants will be randomized to view a fast-food menu featuring one of seven labeling conditions and then will answer questions about the participant's reactions to and interpretations of the label, perceived label effectiveness, intention to purchase a menu item with the label, as well as perceptions of two fast-food menu items.

DETAILED DESCRIPTION:
This survey will explore the perceptions and understanding of different hypothetical menu label designs related to sustainability and environmental harm compared to a control label The survey research firm CloudResearch will recruit a sample of ~12,400 adults aged 18 years and older who reside in the United States.

Participants will be randomized to view a fast-food online ordering menu with one of seven labeling schemes applied: (1) a QR code on all items (control); (2) Low Sustainability labels; (3) Unsustainable labels; (4) Environmental Harm labels; (5) High Environmental Harm labels; (6) High Environmental Cost labels; and (7) numeric Environmental Cost labels on all items. All fast-food menus will include a selection of main entrée items. The control QR code and numeric environmental cost labels will display labels on all menu items. All other label conditions will apply labels only to items with higher environmental impact as defined by ingredient-level environmental impact estimates based on the Cool Food Pledge Calculator.

Participants will be shown the menu and the label in isolation and will then be asked about interpretations of the label, reactions to the label, perceived message effectiveness (PME) of the label, how helpful the participants find the label to be, and the intention to purchase a menu item with the label. The participants will also be shown two different individual fast-food items with the label to which the participants were randomized (if applicable) in random order and asked about the perceived appeal, healthfulness, and environmental impact of the menu items.

The primary outcome in this exploratory study will be intention to purchase a hypothetical menu item with the label shown. Secondary outcomes include label interpretation, perceived label understandability, perceived label believability, perception that the label grabbed attention, perceived message effectiveness (PME) of the label, perceived helpfulness of the label, perceived level of appeal of menu items, perceived level of healthfulness of menu items, and perceived environmental impact of menu items.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Member of the CloudResearch panel
* Residing in the United States

Exclusion Criteria:

* - <18 years of age
* Not residing in the United States
* Completed the survey implausibly quickly based on the distribution of the time to complete the survey among all participants
* Failed the built-in Qualtrics survey fraud detection measures
* Failed the attention check question included in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14720 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Intention to purchase | Immediately after viewing the menu excerpt and label image
  Intention to purchase is measured with the survey question: "How likely would you be to purchase a menu item with this label?" Response options are a 7-point Likert scale: 1=Very unlikely, 2=Unlikely, 3=Somewhat unlikely, 4=Neither likely nor unlikely, 5=Somewhat likely, 6=Likely, 7=Very likely. A higher rating is better.

SECONDARY OUTCOMES:
Label interpretation | Immediately after viewing the menu excerpt
  Label interpretation is assessed with a survey question: "Imagine that you are in a fast-food restaurant (such as Burger King) to order lunch. Next are questions about the label, as displayed on the menu example below. If you saw this label next to an item on the menu, what would you think the label indicates about the item? [check all that apply]". Response options provided are a range of statements about the menu item: 1="This menu item is unhealthy", 2="This menu item is healthy" 3="This menu item is good for the environment", 4="This menu item used a lot of natural resources (e.g. land, water) to produce", 5="This menu item will keep you full for a long time", 6="This menu item is bad for the environment", and 7="This menu item will cost consumers more to purchase". Also included are 8="I don't know" and 9="Other" option with open-text entry.
Perceived label understandability | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label is easy to understand". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived label believability | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label is believable to me". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perception that label grabbed attention | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label grabs my attention". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived message effectiveness (PME) as assessed by the University of North Carolina (UNC)-PME scale | Immediately after viewing the menu excerpt and label image
  Perceived message effectiveness (PME) is measured using the unipolar 3-item University of North Carolina (UNC)-PME scale. Participants will be asked how much each label discourages consumption of or evokes concern of unpleasantness about consumption of foods with the label. After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statements: "This label discourages me from wanting to eat foods with this label", "This label makes foods with this label seem unpleasant", and "This label makes me concerned about the health effects of eating menu items with this label". Response options are a 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived label helpfulness | Immediately after viewing the menu excerpt and label image
  Perceived label helpfulness is measured with the survey question: "How helpful would you find this label when deciding what to order at a fast-food restaurant?" Response options are a 7-point Likert scale: 1=Very unhelpful, 2=Unhelpful, 3=Somewhat unhelpful, 4=Neither helpful nor unhelpful, 5=Somewhat helpful, 6=Helpful, 7=Very helpful. A higher ranking is better.

OTHER OUTCOMES:
Perceived level of appeal of food items | Immediately after viewing each menu item
  Perceived level of appeal of food item is measured after showing participants two different individual menu items separately by label condition. After showing each item, the survey question asks, "How appealing do you think this item is?", and response options are a 7-point Likert scale: 1=Very unappealing, 2=Unappealing, 3=Slightly unappealing, 4=Neither appealing nor unappealing, 5=Slightly appealing, 6=Appealing, 7=Very appealing. A higher ranking is better
Perceived level of healthfulness of food item | Immediately after viewing each menu item
  Perceived level of healthfulness of labeled food item is measured after showing participants two different individual menu items separately by label condition. After showing each item, the survey question asks, "How healthy do you think this item is?", and response options are a 7-point Likert scale:1=Very unhealthy, 2=Unhealthy, 3=Slightly unhealthy, 4=Neither unhealthy nor healthy, 5=Slightly healthy, 6=Healthy, 7=Very healthy. A higher ranking is better.
Perceived level of environmental impact of food item | Immediately after viewing each menu item
  Perceived level of environmental impact of labeled food item is measured after showing participants two different individual menu items separately by label condition. After showing each item, the survey question asks, "What do you think the environmental impact of this item is?", and response options are a 7-point Likert scale:1=Extremely high environmental impact, 2=Very high environmental impact, 3=High environmental impact, 4=Moderate environmental impact, 5=Low environmental impact, 6=Very low environmental impact, 7=Extremely low environmental impact.

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Wolfson, PhD, MPP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share anonymous individual level data with members of the research team and with other interested researchers upon request. After results have been published the investigators will make study data available on Open Science Framework consistent with the Data Sharing and Management Plan.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the study team has published results, the investigators will make data and other documents available. There is no end date for availability.
Access Criteria: Data and supporting documentation will be publicly available on the Open Science Framework website.